CLINICAL TRIAL: NCT01407341
Title: ChronOS Stability Study: For Metastatic Cancer
Brief Title: Beta-Tricalcium Phosphate Bone Graft in Treating Patients Undergoing Surgery For Metastatic Spine Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0S-09-12; NCI-2011-01243 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2012-08

CONDITIONS: Adult Spinal Cord Neoplasm; Spinal Bone Metastases; Spinal Cord Compression
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Cord Compression | interventions — Therapeutics; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (ChronOS) (Experimental): Patients undergo placement of beta-tricalcium phosphate bone graft strips posterolaterally during surgery.
  Interventions: Procedure: musculoskeletal complications management/prevention; Procedure: bone graft; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Procedure: musculoskeletal complications management/prevention — Receive beta tricalcium-phosphate bone graft
  Other Names: complications management/prevention, musculoskeletal; management/prevention, musculoskeletal complications
Procedure: bone graft — Receive beta tricalcium-phosphate bone graft
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies beta-tricalcium phosphate bone graft in treating patients undergoing surgery for metastatic spine cancer. A bone graft may help healing and bone growth in patients undergoing surgery for spine cancer

DETAILED DESCRIPTION:
OBJECTIVES: I. To determine if Chronos (beta-tricalcium phosphate bone graft) will form a posterolateral fusion mass in patients undergoing fusion surgery for spine cancer within 12 months. II. To evaluate quality of life following the use of ChronOS as measured by (a) pain (or lack of pain) associated with pseudoarthrosis and (b) the need for additional treatment for instability as a result of hardware failure. OUTLINE: Patients undergo placement of beta-tricalcium phosphate bone graft strips posterolaterally during surgery. After completion of study treatment, patients are followed up at 1 month and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgery for spinal decompression for tatic spine cancer who require bone substitute for a posterolateral spinal fusion
* Patients may or may not have posterolateral instrumentation

Exclusion Criteria:

* Status-post previous fusion with allogeneic bone graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Achievement of durable posterolateral fusion | Within 12 months
  Measured from x-ray and/or computed tomography (CT) scans. Standard criteria of determining fusion is visualization of continuous trabeculating bone bridging the transverse processes and facets on AP and lateral x-rays or when there is < 2 degree angular motion and < 2mm of translation on standing flexion and extension radiographs.

SECONDARY OUTCOMES:
Achievement of posterolateral fusion | Up to 12 months
Occurrence of subsequent hardware failure | Every 3 months for 12 months
Requirement of additional treatment is for instability | Within 12 months
First documentation of posterolateral fusion | Within 12 months
Occurrence of pain or disability experienced after surgery that is related to spinal metastasis or is a consequence of the resulting treatment | Every 3 months for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chen, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States